CLINICAL TRIAL: NCT02299921
Title: Effect of Alcohol and Drugs of Abuse on Immune Function in Critically Ill Patients With Respiratory Failure
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 14-0630; R24AA019661 (NIH)
Record Dates: First submitted 2014-11-19; First posted 2014-11-24 (Estimated); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Infection; Alcohol Abuse; Drugs of Abuse; Lung Injury
MeSH Terms: conditions — Infections; Alcoholism; Substance-Related Disorders; Lung Injury | interventions — Ethanol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood: serum cortisol, Adrenocorticotropic Hormone (ACTH), Corticotropin-Releasing Hormone (CRH), Arginine Vasopressin (AVP) hair: cortisol urine: Total Protein (TP), Neutrophil Gelatinase-Associated Lipocalin (NGAL), Kidney Injury Molecule-1 (KIM-1) exhaled breath condensate: Chemokine ligand 5 (CCL5) Bronchoalveolar lavage (BAL): cell count and differential, total protein, cytokines/chemokines including CCL5, Tumor Necrosis Factor a (TNFa), Interferon Gamma (IFNg), Interleukin 6 (IL-6), IL-8, IL-10, alveoloar macrophage cytokine/chemokine production, alveolar macrophage viability, apoptosis, cytotoxicity, lymphocyte activation.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adult ICU patients with respiratory problem: Adult medical ICU patients admitted to the University of Colorado Hospital for a primary respiratory problem, and who are expected to require ICU care ≥48 hrs.
  Interventions: Other: Characterize alcohol and drug use
- Intubated Adult ICU patients with respiratory failure: A subset of subjects, adult medical ICU patients with respiratory failure (due to underlying lung pathology) and who require endotracheal intubation and mechanical ventilation.
  Interventions: Other: Characterize alcohol and drug use

INTERVENTIONS:
Other: Characterize alcohol and drug use — Characterize alcohol and drug use in patients newly admitted to the medical ICU service, who are expected to stay in the ICU for greater than 48 hours. The investigators will collect blood, exhaled breath condensate, urine and hair samples over the first 10 days of hospitalization. A select subset of subjects will have bronchoalveolar lavage (BAL) obtained.

SUMMARY:
This study plans to learn more about people who are sick in the hospital with a lung infection, or respiratory failure. Respiratory failure, or severe lung failure, is a life-threatening disease. When it happens, the lungs have trouble carrying out their normal function of getting oxygen into the blood, and removing carbon dioxide from the body. Investigators are conducting this study to see what drinking too much alcohol, using tobacco products, or using drugs (both legal and illegal) may do to lung infections and respiratory failure.

Subjects are asked to be in this research study because they are thought to have a lung infection and may also have respiratory failure. Alcohol, tobacco, and drug use have been linked to lung infections, respiratory failure, and even death, but the reasons for this aren't known. People who use unhealthy amounts of alcohol, tobacco, and or drugs may be more at risk for lung infections, and for severe complications due to lung infection. Subject participation is important whether or not you use alcohol and or drugs.

ELIGIBILITY:
Inclusion criteria:

* Specific Aim 1: Adult medical ICU patients admitted to the University of Colorado Hospital for a primary respiratory problem, and who are expected to require ICU care ≥48 hrs
* Specific Aim 2: (1) Adult medical ICU patients with respiratory failure (due to underlying lung pathology) and who require endotracheal intubation and mechanical ventilation. (2) Adult medical and other ICU patients with respiratory failure, not related to a lung condition, and who require endotracheal intubation and mechanical ventilation. (3) Adult ICU patients previously admitted to the University of Colorado Hospital for a primary respiratory problem, and who required care ≥48 hrs.

Exclusion criteria, Specific Aim 1 and 2:

* Patients who are expected to require ICU care <48 hrs
* Patients admitted to the ICU who are not ICU status (being housed for space issues)
* Patient is unlikely to survive 48 hours
* Patient is on comfort care (hospice measures)
* Patients less than 18 or greater than 90 years of age
* Patient is a prisoner
* ICU attending declines enrollment of patient
* Patients who are pregnant
* Patients who have significant anemia, defined as Hgb<8% or Hct<24%, or who have evidence of active bleeding.

For bronchoscopy portion of Specific Aim 2.

* Patients who are on either a fraction of inspired oxygen inspired oxygen fraction (FiO2)>80% or positive end expiratory pressure (PEEP) >10 cm H20
* Patients with platelets less than 30,000(chronically)
* Patients who are expected to undergo a spontaneous breathing trial within the next 4 hours
* Patients with an order or plan to extubate in the next 4 hours
* Patients who have an endotracheal tube (ETT) <7.5 F
* Patients who are currently dangerously agitated
* Pregnant women

Exclusion criteria (outpatients ONLY for SA2 (3)):

1. Patients who required ICU care <48 hrs
2. Patients less than 18 or greater than 90 years of age
3. Patient is a prisoner
4. Patients who are pregnant
5. Residency > 40 miles from UCH clinics
6. non-English or non-Spanish speaking
7. Inability to perform study procedures (i.e. physical disability)
8. unable to perform pulmonary function testing
9. diagnosis of chronic pulmonary disease (e.g. COPD)
10. diagnosis of chronic neurodegenerative disease or severe dementia
11. history of anoxic or traumatic brain injury
12. prior ICU hospitalization at a non-UCH facility.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Specific Aim 1. Adult medical ICU patients admitted to the University of Colorado Hospital for a primary respiratory problem, and who are expected to require ICU care ≥48 hrs
  Specific Aim 2. Adult medical ICU patients with respiratory failure (due to underlying lung pathology) and who require endotracheal intubation and mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-11 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of alcohol use disorders (AUDs) | prevalence, absolute value and change over 7 days, 3 Month follow up, 6 Month follow up
  Among medical ICU (MICU) patients who remain in ICU greater than or equal to 48 hours: Prevalence of alcohol use disorders (AUDs), drug use disorders (DUDs), their combination (both), or no AUD/DUDs. Absolute value, and change over 7 days, in serum/urine/exhaled breath condensate/hair cortisol, corticotropin releasing hormone (CRH), adenovirus proteinase (AVP), and adrenocorticotropic hormone (ACTH), stratified by AUD/DUD/both/neither. 3 Month and 6 Month follow up were added to this outcome measure via a protocol amendment after study-start.
Incidence and etiology of respiratory failure, stratified by AUD/DUD/both/neither | participants will be followed for the duration of hospital stay, an expected average of 17 days
  Among medical ICU (MICU) patients who develop respiratory failure: Incidence and etiology of respiratory failure, stratified by AUD/DUD/both/neither. Length of time on mechanical ventilation stratified by AUD/DUD/both/neither. Inflammatory profile of BAL stratified by AUD/DUD/both/neither: BAL cell count and differential, Pro-inflammatory BAL cytokines; CCL5, TNFa, interferon-gamma (IFNg), interleukin (IL-1b), interleukin (IL-6). Evidence of oxidative stress in BAL (GSH/glutathione disulfide (GSSG) ratio, pH). Alveolar macrophage activation, degree of apoptosis, and inflammatory cytokine production. Confirm in non-invasively collected samples. Development of Acute Respiratory Distress Syndrome (ARDS) stratified by AUD/DUD/both/neither; Berlin criteria, Lung injury score.
Incidence and etiology of respiratory failure, stratified by AUD/DUD/both/neither: Month 3 | 3 Month follow up
  Among medical ICU (MICU) patients who develop respiratory failure: Incidence and etiology of respiratory failure, stratified by AUD/DUD/both/neither. Length of time on mechanical ventilation stratified by AUD/DUD/both/neither. Inflammatory profile of BAL stratified by AUD/DUD/both/neither: BAL cell count and differential, Pro-inflammatory BAL cytokines; CCL5, TNFa, interferon-gamma (IFNg), interleukin (IL-1b), interleukin (IL-6). Evidence of oxidative stress in BAL (GSH/glutathione disulfide (GSSG) ratio, pH). Alveolar macrophage activation, degree of apoptosis, and inflammatory cytokine production. Confirm in non-invasively collected samples. Development of Acute Respiratory Distress Syndrome (ARDS) stratified by AUD/DUD/both/neither; Berlin criteria, Lung injury score. 3 Month and 6 Month follow up were added to this outcome measure via a protocol amendment after study-start.
Incidence and etiology of respiratory failure, stratified by AUD/DUD/both/neither: Month 6 | 6 Month follow up
  Among medical ICU (MICU) patients who develop respiratory failure: Incidence and etiology of respiratory failure, stratified by AUD/DUD/both/neither. Length of time on mechanical ventilation stratified by AUD/DUD/both/neither. Inflammatory profile of BAL stratified by AUD/DUD/both/neither: BAL cell count and differential, Pro-inflammatory BAL cytokines; CCL5, TNFa, interferon-gamma (IFNg), interleukin (IL-1b), interleukin (IL-6). Evidence of oxidative stress in BAL (GSH/glutathione disulfide (GSSG) ratio, pH). Alveolar macrophage activation, degree of apoptosis, and inflammatory cytokine production. Confirm in non-invasively collected samples. Development of Acute Respiratory Distress Syndrome (ARDS) stratified by AUD/DUD/both/neither; Berlin criteria, Lung injury score. 3 Month and 6 Month follow up were added to this outcome measure via a protocol amendment after study-start.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen L Burnham, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No